CLINICAL TRIAL: NCT02533492
Title: Compare the Results of Antimicrobial to Conventional Suture Materials in Patients Receiving Primary Total Knee Replacement: A Prospective Double-blinded Randomized Controlled Trial
Brief Title: Compare Antimicrobial to Conventional Suture in Patients Receiving Primary Total Knee Replacement
Acronym: Vicryl-Plus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mel Shiuann-Sheng Lee (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Mel Shiuann-Sheng Lee, Chang Gung Memorial Hospital, Dept Orthopedic Surgery, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 98-2933a3
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Wound Infection
Keywords: total knee replacement; vicryl plus; surgical site infection
MeSH Terms: conditions — Wound Infection; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vicryl (Active Comparator): Vicryl suture for wound closure after total knee replacement
  Interventions: Device: vicryl
- vicryl plus (Experimental): Vicryl plus suture for wound closure after total knee replacement
  Interventions: Device: Vicryl plus

INTERVENTIONS:
Device: vicryl — wound closure with vicryl suture
  Other Names: polyglactin
  Arms: Vicryl
Device: Vicryl plus — wound closure with vicryl plus suture
  Other Names: triclosan-coated polyglactin
  Arms: vicryl plus

SUMMARY:
Total knee replacement is now one of the most popular reconstructive procedures for the elderly people to regain their functional capacity and life quality. However the reported incidence of postoperative infection or surgical site infection after total knee replacement has been around 1 to 2 percent. The cost and expenditure for treating periprosthetic infection are high and the results are often detrimental to the patients who suffered from the complication. To decrease the wound healing complication related to the contamination of bacteria, an antibacterial suture was used successfully in some clinical settings and in animal experiments. Whether the antibacterial suture material could be used in patients with total knee replacement has not been addressed in the past. The investigators therefore propose a prospective randomized double-blinded study to investigate the efficacy of an antibacterial suture material in total knee replacement. The inclusion criteria are patients with degenerative osteoarthritis without previous surgery to the index knee. Patients who have inflammatory arthritis such as rheumatoid arthritis, who have neurovascular disease of the lower extremities, who have history of liver cirrhosis or under hemodialysis for renal failure are excluded. One hundred and two patients will be randomized to study group (51 knees) and control group (51 knees) in a period of 12 months. All cases will follow the standard protocol based on clinical pathway. Antibacterial suture material (Vicryl Plus, Ethicon) will be used in the study group and regular suture material (Vicryl, Ethicon) will be used in the control group. Preoperatively, the skin condition (digital photo and image analysis),laser Doppler study, inflammatory markers (CRP/ESR/IL-6), functional score (KSS: Knee Society Score; SF-12: Short Form 12), and VAS score will be assessed. Operative data of operation time, blood loss and wound classification are recorded. Postoperatively, the skin condition (digital photo and image analysis), skin temperature, inflammatory markers, KSS, and VAS will be assessed on 1st and 3rd postoperative day, 2 weeks, 4 weeks, and 3 months.

DETAILED DESCRIPTION:
Title of study:

Compare the results of Antimicrobial with Conventional suture materials in patients receiving primary total knee replacement: a prospective double-blinded randomized controlled trial

Objectives:

Primary Objective: To investigate whether the surgical site infection rate after total knee replacement will be different with two different suture materials.

Secondary Objective: To investigate the surrogating markers for inflammatory response and functional outcomes with two different suture materials.

Rationale:

The reported rate of deep infection following contemporary total knee replacement has been about two percent. The prevalence of prolonged wound drainage of soft tissue complications is between 17 to 50% of patients in whom 1.3% of them eventually developed culture-proved prosthetic infection. Total knee infections typically require complete removal of the prosthesis and prolonged antibiotic treatment. Re-infection rate following revision surgery for infected total knee cases is also significantly higher than those without infection complications. Total knee infections are devastating and associated with prolonged hospital stays, increased co-morbidity, and utilization of medical resources. Measures to reduce the infection rate extensively implemented clinically. However the use of antibacterial suture materials to reduce the wound complications has not yet been investigated before. Clinical trials including this issue only had been discussed in animal studies for minimal series. The effectiveness of the new material should be checked.

This study is designed to investigate the wound conditions and deep infection incidence following total knee replacement performed using either antimicrobial or conventional sutures. A prospective, double-blinded, randomized controlled trial with 102 patients evenly distributed into two groups is proposed. Each group has 51 patients scheduled for unilateral total knee replacement. Randomization is by envelope-drawing to minimize confounding risk factors. One hundred and two sets of suture materials (51 sets of Vicryl Plus and 51 sets of Vicryl) will be separately put into sealed envelopes. The envelopes are randomly assigned with consecutive numbers from 1 to 102. The envelopes are randomly given to the patients for wound closure. Finally, one group of patients will receive antibacterial sutures (VICRYL Plus, Ethicon, Johnson and Johnson, Taipei, Taiwan) following total knee replacement for the wound closure and the other group of patients will receive conventional sutures (VICRYL, Ethicon, Johnson and Johnson, Taipei, Taiwan) following total knee replacement for the wound closure. Group sample sizes of 51 and 51 achieve 81% power to detect a difference of -4% between the null hypothesis that both group means are 9.0 and the alternative hypothesis that the mean is 13.0 with estimated group standard deviations of 6.0 and 8.0 and with a significance level (alpha) of 0.05 using a two-sided two-sample t-test. The primary outcome measure is the incidence of prosthetic infection within three months of surgery. The secondary outcome measures include hospital stay, duration of antibiotics use, pain scale (VAS), wound conditions (wound drainage, extent of erythema, local heat, temperature), and serum parameters during hospitalization and within three months after operation.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative osteoarthritis
* Any age
* Varus/valgus deformity knee

Exclusion Criteria:

* Inflammatory arthritis
* Systemic diseases with coagulopathy
* Immune compromise(ESRD, liver cirrhosis)
* PAOD or DVT history
* Pre-OP INR >1.5
* ASA score >3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
wound infection | 3 months

SECONDARY OUTCOMES:
serum inflammatory marker | 3 months
  ESR, CRP, interleukin-6

OTHER OUTCOMES:
Physiological parameter (skin temperature) | 3 months
  skin temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kweishan, Taoyuan, Taiwan

REFERENCES:
- [Background] Rozzelle CJ, Leonardo J, Li V. Antimicrobial suture wound closure for cerebrospinal fluid shunt surgery: a prospective, double-blinded, randomized controlled trial. J Neurosurg Pediatr. 2008 Aug;2(2):111-7. doi: 10.3171/PED/2008/2/8/111. PMID 18671615
- [Derived] Lin SJ, Chang FC, Huang TW, Peng KT, Shih HN, Lee MS. Temporal Change of Interleukin-6, C-Reactive Protein, and Skin Temperature after Total Knee Arthroplasty Using Triclosan-Coated Sutures. Biomed Res Int. 2018 Jan 15;2018:9136208. doi: 10.1155/2018/9136208. eCollection 2018. PMID 29568771